CLINICAL TRIAL: NCT01321021
Title: Influence of Losartan and Diphenhydramine on Emotional and Cognitive Functions in Healthy Human Subjects
Acronym: LoDi-Basel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dominique de Quervain, MD (Other)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, Prof., MD, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2011DR2032
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Memory, Long-Term; Memory, Short-Term
MeSH Terms: interventions — Losartan; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Losartan, Diphenhydramine, Placebo (Experimental): placebo controlled crossover study with two arms: Losartan, Diphenhydramine
  Interventions: Drug: Losartan, Diphenhydramine, Placebo

INTERVENTIONS:
Drug: Losartan, Diphenhydramine, Placebo — placebo controlled crossover study with two arms: Losartan 40mg, Diphenhydramine 40mg

SUMMARY:
This project aims at identifying novel pharmacological targets for the treatment of memory disorders.

DETAILED DESCRIPTION:
To investigate the effects of the histamine H1 receptor antagonist diphenhydramine and the angiotensin II receptor antagonist losartan on emotional and cognitive functions in healthy human subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* native or fluent German-speaking
* BMI between 19 and 27 kg/m2
* able and willing to give written informed consent and comply with the requirements of the study protocol
* willing to donate saliva sample for DNA-analysis
* female: willing to perform a pregnancy test at the beginning of both test visits

Exclusion Criteria:

* acute or chronic psychiatric or somatic disorder
* pathological ECG
* known hypersensitivity to the IMP under investigation (losartan, diphenhydramine)
* hypotension (RR < 110/70 mmHg)
* bradycardia (< 50 bpm)
* pregnancy, breast-feeding
* long-term medication within last 3 months (oral contraceptives are disregarded)
* smoking (> 3 cigarettes per day)
* concurrent participation in another study
* participation in one of our previous studies using the same memory tests
* inability to read and understand the participant's information

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measures | during cognitive testing at study days
  Memory functions

SECONDARY OUTCOMES:
Secondary Outcome Measures | during cognitive testing at study days
  sleepiness, mood, anxiety, attention, fluid intelligence

CONTACTS AND LOCATIONS:
Overall Officials: Dominique de Quervain, Prof. MD, Principal Investigator — University of Basel, Faculty of Psychology and Medecine, Division of Cognitive Neuroscience
Locations (1):
- University of Basel, Division of Cognitive Neuroscience, Basel, Basel, Switzerland